CLINICAL TRIAL: NCT04312503
Title: Observational Study on the Effect of Switch to Lurasidone or Other Antipsychothics on Metabolic and Weight Changes in Subjects With Schizophrenia"
Brief Title: Observational Study on the Effect of Switch to Lurasidone in Subjects With Schizophrenia"
Acronym: SWITCH
Status: Completed | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Responsible Party: Sponsor
Other Study IDs: 151(A)PO18531
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; lurasidone; antipsychotics; metabolic syndrome; switch
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome | interventions — Lurasidone Hydrochloride; Aripiprazole; Olanzapine; Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COHORT A: Lurasidone: Patients treated with Lurasidone
  Interventions: Drug: Lurasidone
- COHORT B: aripiprazole, olanzapine, quetiapine or risperidone): Patients treated with other atipical antypsicothic as aripiprazole, olanzapine, quetiapine or risperidone)
  Interventions: Drug: aripiprazole, olanzapine, quetiapine or risperidone

INTERVENTIONS:
Drug: Lurasidone — Patients are treated with dosages according clinical practice
  Other Names: Latuda
  Groups: COHORT A: Lurasidone
Drug: aripiprazole, olanzapine, quetiapine or risperidone — Patients are treated with dosages according clinical practice
  Groups: COHORT B: aripiprazole, olanzapine, quetiapine or risperidone)

SUMMARY:
The aim of this study is observation, in an Italian real-world setting, of metabolic effects in patients with schizophrenia who will switch from any mono-therapy or poly-therapy antipsychotic regimen to monotherapy with lurasidone or to one of the other four most used atypical antipsychotics.

DETAILED DESCRIPTION:
The aim of this study is the observation, in psychiatric Italian real-world settings, of metabolic effects, effectiveness, side effects and therapeutic adherence in patients with schizophrenia who switched, for any reason (efficacy, safety, metabolic problems, therapeutic adherence or patient's request), from any mono-therapy or poly-therapy antipsychotic regimen to monotherapy with lurasidone or with one of the four most used atypical antipsychotics in Italy (aripiprazole, olanzapine, quetiapine, risperidone). Patient's past medical and psychiatric history of the last 12 months will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia according to DSM-5.
* Patients who gave their written consent for participation in the study and for personal data processing and willing to comply with all study procedures.
* Male and female patients ≥ of 18 years old at baseline.
* Patients treated or in treatment with any typical or atypical antipsychotic monotherapy or polytherapy.
* Patients switched from the pre-existing therapy to lurasidone, aripiprazole, olanzapine, quetiapine or risperidone in monotherapy within the preceding 2 weeks. The date of the switch is considered as baseline.

Exclusion Criteria:

* Female patients who are pregnant or lactating
* Patients fulfilling DSM-5 criteria for diagnosis of bipolar disorder and/or dementia.
* Amphetamines and/or Opiates abuse or dependence , as defined by DSM-5 criteria.
* Patients with no history of antipsychotics use.
* Patients recruited in another study as follows:
* currently enrolled in any pharmacological or non-pharmacological, interventional or observational study:
* who participated in the last 30 days to any observational or no-profit interventional study;
* who participated in the last 12 months to any interventional commercially sponsored study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients (aged > 18 years) affected by schizophrenia according to DSM-5 (Appendix A).
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in the metabolic parameters | 4 weeks
  Change in metabolic syndrome in 3 of 5 parameters:
  1. Arterial hypertension defined as. systolic pressure ≥ 130 mmHg and/or diastolic pressure ≥85 mmHg or treatment for hypertension.
  2. Waist Circumference ≥ 90 cm in men or ≥ 80 cm in women.
  3. Fasting Plasma Glucose ≥5.6 mmol/l and/or known treatment for hyperglycemia.
  4. Triglycerides ≥1.7 mmol/l or medication for elevated triglycerides.
  5. HDL Cholesterol ≤ 1.0 mmol/l in men and ≤1.3 mmol/l for women or taking medication.

SECONDARY OUTCOMES:
Retrospective investigation of the metabolic effects of switches to any atypical antipsychotic occurred in the previous 12 months | 12 months before baseline (switch to any atypical antipsychotics)
  Change in metabolic syndrome in 3 of 5 parameters:
  1. Arterial hypertension defined as. systolic pressure ≥ 130 mmHg and/or diastolic pressure ≥85 mmHg or treatment for hypertension.
  2. Waist Circumference ≥ 90 cm in men or ≥ 80 cm in women.
  3. Fasting Plasma Glucose ≥5.6 mmol/l and/or known treatment for hyperglycemia.
  4. Triglycerides ≥1.7 mmol/l or medication for elevated triglycerides.
  5. HDL Cholesterol ≤ 1.0 mmol/l in men and ≤1.3 mmol/l for women or taking medication.

CONTACTS AND LOCATIONS:
Locations (18):
- Italy (18):
  - Ospedali Riuniti SOD di Clinica Psichiatrica, Ancona, AN
  - Spedali Civili di Brescia Dipartimento di Salute Mentale 1, Brescia, BS
  - A.O.U. di Cagliari Corso Vittorio Emanuele II, 6 09124 Cagliari (CA), Cagliari, CA
  - P.O. Gaspare Rodolico - U.O.C. di Psichiatria, Catania, CT
  - AO Mater Domini U.O. Psichiatria, Catanzaro, CZ
  - A.O.U. Ospedali Riuniti di Foggia - S.P.D.C. Viale Pinto 71121 Foggia (FO), Foggia, FG
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - DSM Dipartimento Salute Mentale, Lecce, LE
  - Ospedale S. Gerardo Università Bicocca Dipartimento di Salute Mentale, Monza, MB
  - Ospedale Maggiore Policlinico di Milano U.O. C. di Psichiatria, Milan, MI
  - Ospedale San Raffaele U.O.C. Psichiatria Generale e Riabilitazione, Milan, MI
  - Ospedale Luigi Sacco, S.C. Psichiatria 2, Milan, MI
  - III S.P.D.C. Azienda Ospedaliera di Padova 35128 Padova - (PD), Padua, PD
  - Clinica Von Sibenthal Via della Madonnina, 1, Genzano di Roma, RM
  - Azienda Ospedaliero Universitaria Sant'Andrea, Roma, RM
  - A.O.U. San Luigi Gonzaga - S.C.D.U. di Psichiatria Regione Gonzole, 10, Orbassano, TO
  - Azienda Ospedaliera Universitaria Federico II - U.O. Psichiatria, Napoli
  - Azienda Ospedaliera - Universitaria Senese, Siena